CLINICAL TRIAL: NCT00795470
Title: A Pilot Concealed Randomized Double-blinded Placebo-controlled Factorial Trial of Antimicrobial Therapy and/or Catheter Change for Catheter-associated Urinary Tract Infections in the Critically Ill
Brief Title: Factorial Trial of Antimicrobial Therapy and/or Catheter Change for Catheter Urinary Tract Infections.
Acronym: CAUTION
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Not pursuing the study due to funding issues
Sponsor: Unity Health Toronto (Other)
Collaborators: Kingston Health Sciences Centre (Other); Mount Sinai Hospital, New York (Other); The Ottawa Hospital (Other); Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REB 08-287
Record Dates: First submitted 2008-11-20; First posted 2008-11-21 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-11

CONDITIONS: Urinary Tract Infections
Keywords: urinary tract infection; critically ill; ICU; antimicrobial; Catheter associated urinary tract infections
MeSH Terms: conditions — Urinary Tract Infections; Critical Illness | interventions — Anti-Infective Agents

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- No catheter change no antimicrobial (No Intervention): Urinary catheter will not be changed and no antimicrobials will be prescribed
- Antimicrobial and catheter change (Active Comparator)
  Interventions: Drug: Antimicrobial; Device: Catheter change
- Catheter change and NO antimicrobial (Active Comparator)
  Interventions: Device: Catheter change
- Antimicrobial and NO catheter change (Active Comparator)
  Interventions: Drug: Antimicrobial

INTERVENTIONS:
Drug: Antimicrobial — Appropriate antimicrobial based on urine culture results
  Arms: Antimicrobial and NO catheter change; Antimicrobial and catheter change
Device: Catheter change — Change urine catheter
  Arms: Antimicrobial and catheter change; Catheter change and NO antimicrobial

SUMMARY:
Urinary tract infection (UTI) is a common infection in patients in the intensive care unit (ICU) that increases length of stay but not mortality. It is not known whether antibiotic treatment will alter outcomes. Our previous studies have documented wide practice variations exist amongst doctors, including prescribing antibiotics to asymptomatic patients. Therefore, the merits of various ways to manage the infection require further studies to minimize the potential for over-prescribing of antibiotics, a practice that can increase the development of resistant bacteria.

The objective of this pilot study is to determine the feasibility of conducting a larger definitive study that will determine the effect of catheter change and/or systemic antibiotics as compared to no interventions on outcomes and resource utilization in ICU patients with UTI. Patients will be randomized to receive no treatment, antibiotics alone, urine catheter change alone, and both catheter change and antibiotics. Their clinical outcomes will be assessed.

Results from the pilot trial will provide information about whether it is feasible to conduct the larger definitive trial. Results of the definitive study will provide guidance to clinicians on how to manage a frequent clinical problem and optimize antibiotic usage.

ELIGIBILITY:
Inclusion Criteria:

1. Adult ICU patient (≥ 18 years old)
2. Admitted to the ICU for ≥ 96 hours
3. Indwelling urinary catheter in place for ≥ 48hours that was inserted during this hospital admission
4. Urine culture positive (≥ 105 CFU/mL) for 1 or 2 organism (s) (e.g. bacteria or fungus)
5. Have received antimicrobial therapy that would cover the isolated organism(s) in the index urine culture for < 24 hours (i.e. therapy that does NOT cover the isolated organism(s) in the index urine culture of any duration or antimicrobial that covers the index urine organism for < 24 hours are permitted)

Exclusion Criteria:

1. Suspected or confirmed pyelonephritis, renal abscess, or concurrent bacteremia with the same organism(s) as those isolated in the index urine culture
2. Anuria (< 50 mL/day)
3. Imminent death within 48 hours or decision to withdraw supportive care by clinical team
4. Neutropenia (< 500/mm3)
5. Patient has an alternative infection and requires an antimicrobial that has a spectrum of activity which include all the organism(s) isolated from the index urine culture
6. Mixed fungal/bacterial CAUTI (i.e. index urine culture contains both bacteria and fungus)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Number of patients enrolled | 18 months
  none enrolled
Protocol Adherence Rate | 18 months

SECONDARY OUTCOMES:
ICU free days at Day 30 | 30 days
Microbiologic Outcome | Day 7 and 14
Developement of resistance | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Jan Friedrich, DPhil, MD, MSc, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Chant C, Dos Santos CC, Saccucci P, Smith OM, Marshall JC, Friedrich JO. Discordance between perception and treatment practices associated with intensive care unit-acquired bacteriuria and funguria: a Canadian physician survey. Crit Care Med. 2008 Apr;36(4):1158-67. doi: 10.1097/CCM.0b013e3181692af9. PMID 18379242